CLINICAL TRIAL: NCT06175130
Title: Cross-sectional Dietary Intake Survey on Ivorian School-aged Children (6-12 yo) and Women of Reproductive Age (15-50 yo)
Brief Title: Cross-sectional Dietary Intake Survey on Ivorian School-Aged Children and Women of Reproductive Age
Acronym: AN
Status: Completed | Type: Observational
Sponsor: FrieslandCampina (Industry)
Collaborators: Société de Nutrition de Côte d'Ivoire (Unknown)
Responsible Party: Sponsor
Other Study IDs: AfricaNutrition
Record Dates: First submitted 2023-11-28; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diet; Deficiency
Keywords: Nutrient Inadequacy; Dietary Patterns; Food Intake
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy children (6-12 years): Healthy children (6-12 years), no illness or disease
- Healthy Women of reproductive age (15-50 years): Healthy Women of reproductive age (15-50 years), no illness or disease

SUMMARY:
A cross-sectional dietary intake study was conducted with 423 Ivorian school aged children (SAC, 6-12 years) and 423 women of reproductive age (WRA, 15-49 years) from four cities, recruited by two-stage random sampling.

DETAILED DESCRIPTION:
A cross-sectional dietary intake study was conducted with 423 Ivorian school aged children (SAC, 6-12 years) and 423 women of reproductive age (WRA, 15-49 years) from four cities, recruited by two-stage random sampling. Dietary intake data were collected by multiple pass 24-hour recall. For a sub-sample (10% subjects) two-day non-consecutive multiple pass 24-hour recall was collected.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* illness or disease

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: healthy children and women living in the cities of Ivory Coast
Sampling Method: Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mean usual nutrient intake per day | Standard multiple pass 24-hour recall
  Mean usual nutrient intake of iron (mg), zinc (mg), vitamin A (RAE), calcium(mg), vitamin B1 (g), B2 (mg), B3 (mg), B6 (mg), B9 (ug), B12 (ug) and vitamin D (ug DFE) will be calculated based on food intake per person per day conversion to usual nutrient intakes per person per day using food composition tables.

SECONDARY OUTCOMES:
Nutritional status (Prevalence of stunting, underweight, overweight and obesity) | on the spot measurement
  Height and weight were measured using standardized scales and height boards. Calculations were made comparing the individual's weight, height and age in some cases to define nutritional status indicators. Cut-offs used were defined by World Health Organization (WHO) Anthro Plus Software (version 1.0.4) for children and using WHO cut-off values for adults. Underweight (<18.5 kg/m2), normal (18.5-24.9 kg/m2), overweight (25-29.9 kg/m2) and obese (>30 kg/m2).
Food intake per day per person | Standard multiple pass 24-hour recall
  Food item and food group intake will be calculated based on classification of foods consumed into food groups

CONTACTS AND LOCATIONS:
Locations (1):
- FrieslandCampina Research and Development, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared

REFERENCES:
- [Derived] Ayling K, Talsma EF, Konan AG, Tiahou G, Gbane M, Bovee-Oudenhoven I, Melse-Boonstra A. Assuming the "Best-Fit" Shape of the Usual Nutrient Intake Distribution (with nutriR) Does Not Affect Prevalence Estimates of Nutrient Intake Inadequacy: Results from a Dietary Intake Survey in Ivorian School-Age Children. J Nutr. 2025 Jul;155(7):2449-2458. doi: 10.1016/j.tjnut.2025.05.023. Epub 2025 May 23. PMID 40414299